CLINICAL TRIAL: NCT01211444
Title: US Prospective Clinical Study of the Apnex Medical Hypoglossal Nerve Stimulation (HGNS) System to Treat Obstructive Sleep Apnea
Brief Title: US Clinical Study of the Apnex Medical Hypoglossal Nerve Stimulation (HGNS) System to Treat Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Apnex Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-004
Record Dates: First submitted 2010-08-20; First posted 2010-09-29 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2011-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; OSA; Hypoglossal nerve stimulation; Sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HGNS System (Experimental)
  Interventions: Device: HGNS Treatment

INTERVENTIONS:
Device: HGNS Treatment — The Apnex Hypoglossal Nerve Stimulation System (HGNS) is an implanted medical device that is designed to prevent the tongue from blocking the airway during sleep. It is fully automatic and can be implanted during a simple surgical procedure. After it is implanted, the device is programmed to meet the unique needs of each patient. The device is on when the patient is sleeping and off when the patient is awake.

SUMMARY:
The overall goal of the study is to evaluate the safety, efficacy and therapy settings of the Hypoglossal Nerve Stimulation (HGNS) System for stimulating the hypoglossal nerve to help maintain airway opening in subjects with Obstructive Sleep Apnea (OSA).

ELIGIBILITY:
Eligibility Criteria

1. Previously diagnosed with moderate-to-severe obstructive sleep apnea.
2. Subject has failed or does not tolerate CPAP treatment.
3. Age between 21 and 70 years.
4. Body mass index (BMI) less than or equal to 37.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mean change in AHI measured with in-lab nighttime polysomnography (PSG) compared to baseline | 6 months post-implant
Mean change in functional outcomes measured with the Functional Outcomes Sleep Questionnaire (FOSQ) compared to baseline | 6 months post-implant
The frequency of serious adverse events. | One month post-implant.
The frequency of serious adverse events. | 3 months post-implant.
The frequency of serious adverse events. | 6 months post-implant.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Freeman, PhD, Principal Investigator — Clinilabs, Inc. West Side ENT, NY, NY; Tod Huntley, MD, Principal Investigator — Center for Ear, Nose, Throat and Allegery, PC (Centa), Carmel, IN; Con Iber, MD, Principal Investigator — Dept of Neurology, University of Minnesota; Eric Kezirian, MD, Principal Investigator — University of Califoprnia - San Francisco
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Saint Vincent Hospital, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Clinilabs, Inc., New York, New York

REFERENCES:
- See also: Related Info — http://www.apnexmedical.com